CLINICAL TRIAL: NCT06277908
Title: 90-day Postoperative Morbidity and Mortality After Elective Surgery for Gastric Cancer
Brief Title: Postoperative Morbidity and Mortality After Gastric Cancer Surgery
Acronym: GASTROSTAT
Status: Not yet recruiting | Type: Observational
Sponsor: P. Herzen Moscow Oncology Research Institute (Other Government)
Collaborators: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Andrey Ryabov, Head of Department of Thoracoabdominal Oncology, P. Herzen Moscow Oncology Research Institute
Other Study IDs: 110-1
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer; Siewert Type III Adenocarcinoma of Esophagogastric Junction; Stomach Cancer
Keywords: Gastric cancer; Surgery; Morbidity; Mortality
MeSH Terms: conditions — Stomach Neoplasms | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with morbidity: Patients who suffered from any type of morbidity after surgery
  Interventions: Procedure: Elective Surgery for gastric cancer
- Patients without morbidity: Patients who did not suffer from any type of morbidity after surgery
  Interventions: Procedure: Elective Surgery for gastric cancer

INTERVENTIONS:
Procedure: Elective Surgery for gastric cancer — Total, distal or proximal gastrectomy via open, laparoscopic or robotic approach

SUMMARY:
Gastric cancer is still one of the main health care issue and gastrectomy with lymph node dissection is the only chance to be cure. Trials show that the postoperative course differs significantly between eastern and western centers, as well as between clinics within Russian Federation. Postoperative 30-day postoperative mortality after gastric cancer surgery ranges from 1% to 5%, and postoperative complication rates range from 10% to 40%. To improve the quality of further studies and recommendations for standardization of surgical treatment of gastric cancer and its complications, there is a need to study the differences in 90-day postoperative morbidity and mortality in different clinics and centers of the Russian Federation.

DETAILED DESCRIPTION:
According to 2018 World Health Organization (WHO) data, gastric cancer is the fourth most common malignant disease and the third leading cause of cancer-related deaths worldwide. Surgery with lymphadenectomy remains the standard of care. Despite significant changes in gastric cancer treatment protocols, surgery is still associated with high risks of complications, with rates varying from clinic to clinic. And currently, the use of multimodal treatments and standardization of surgical procedures are proposed as strategies to improve outcomes. In addition, the use of laparoscopic and robotic techniques have been proposed to provide better short-term results compared to open surgery and comparable long-term oncological outcomes. Randomized trials show that the postoperative course differs significantly between eastern and western centers, as well as between clinics within Russian Federation. Postoperative 30-day postoperative mortality after gastric cancer surgery ranges from 1% to 5%, and postoperative complication rates range from 10% to 40%. While mortality is easier to quantify, there are no standardized criteria for calculating postoperative complication rates. To improve the quality of further studies and recommendations for standardization of surgical treatment of gastric cancer and its complications, there is a need to study the differences in 90-day postoperative morbidity and mortality in different clinics and centers of the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with primary gastric malignancy (including Siewert III) undergoing elective surgery with curative intent (either total or partial gastrectomy) via open, laparoscopic or robotic approach between 18th March 2024 and 18th September 2024.

Exclusion Criteria:

* Patients with clinical evidence of metastatic disease, including positive peritoneal cytology on previous staging laparoscopy,
* Patients with known synchronous cancer;
* Patients with Gastrointestinal stromal tumors (GIST)
* Presence of gastroesophageal junction (Siewert I and II) malignancy;
* Patients submitted to Emergency surgery or surgery without curative intent;
* Patients undergoing additional surgery (except cholecystectomy) along with surgery for gastric cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with primary gastric malignancy (including Siewert III) undergoing elective surgery with curative intent (either total or partial gastrectomy) via open, laparoscopic or robotic approach between 18th March 2024 and 18th September 2024.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the type of complications and the incidence of it | within 90 days after operation
  the types of complication is classified into as follows: anastomotic leak, postoperative bleeding requiring invasive treatment, other complications requiring re-intervention or other invasive procedure, postoperative bowel obstruction, postoperative pancreatic fistula, duodenal leak, gastrostasis, postoperative pancreatitis, postoperative bowel perforation or necrosis, non-surgical infections, pleural effusion requiring drainage, respiratory failure requiring reintubation, acute renal failure requiring hemofiltration/dialysis, need for prolonged intubation, need for tracheostomy, need for cardiopulmonary resuscitation, pulmonary embolism, pneumothorax requiring treatment, myocardial infarction, acute myocardial failure, cardiac dysrhythmia requiring invasive treatment, stroke, acute liver dysfunction, other complications.
  Each complication will be graded according to Clavien-Dindo classification. Re-admission or visiting emergency room will be checked and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Ryabov, MD, PhD, Study Director — P.Herzen Moscow Oncological Research Institute; Vladimir Khomyakov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Nuriddin Abdulkhakimov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Pavel Smirnov, Principal Investigator — P.Herzen Moscow Oncological Research Institute
Locations (9):
- Russia (9):
  - A.S. Loginov Moscow Clinical Scientific Center, Moscow
  - A.Tsyb Medical Radiological Research Centre, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - P.Herzen Moscow Oncological Research Institute, Moscow
  - Petrovsky National Research Centre of Surgery, Moscow
  - Vishnevsky National Medical Research Center of Surgery, Moscow
  - Nizhny Novgorod Regional Clinical Oncological Dispensary, Nizhny Novgorod
  - National Medical Research Centre for Oncology, Rostov-on-Don
  - Petrov National Medical Research Center of Oncology, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided